CLINICAL TRIAL: NCT00684801
Title: Improving the Quality of Advanced Cancer Care With Disease Management
Brief Title: Disease Management Program or Usual Care in Patients With Stage III or Stage IV Lung Cancer, Pancreatic Cancer, Ovarian Cancer, or Colorectal Cancer, and Their Caregivers
Status: Completed | Type: Observational
Sponsor: Case Comprehensive Cancer Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Other Study IDs: CASE6Y07; P30CA043703 (NIH); CASE6Y07 (Other: Case Comprehensive Cancer Center); CASE-6Y07-CC333 (Other: Cancer Center IRB)
Record Dates: First submitted 2008-05-23; First posted 2008-05-28 (Estimated); Last update posted 2015-10-09 (Estimated); Status verified 2015-10

CONDITIONS: Colorectal Cancer; Lung Cancer; Ovarian Cancer; Pancreatic Cancer
Keywords: recurrent non-small cell lung cancer; recurrent small cell lung cancer; stage IIIA non-small cell lung cancer; stage IIIB non-small cell lung cancer; stage IV non-small cell lung cancer; extensive stage small cell lung cancer; recurrent pancreatic cancer; stage III pancreatic cancer; stage IV pancreatic cancer; recurrent ovarian epithelial cancer; recurrent ovarian germ cell tumor; stage III ovarian epithelial cancer; stage III ovarian germ cell tumor; stage IV ovarian epithelial cancer; stage IV ovarian germ cell tumor; recurrent colon cancer; stage III colon cancer; stage IV colon cancer; recurrent rectal cancer; stage III rectal cancer; stage IV rectal cancer
MeSH Terms: conditions — Colorectal Neoplasms; Lung Neoplasms; Ovarian Neoplasms; Pancreatic Neoplasms; Carcinoma, Non-Small-Cell Lung; Small Cell Lung Carcinoma; Carcinoma, Ovarian Epithelial; Colonic Neoplasms; Rectal Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (2):
- Usual care (control group): Patients undergo usual care as determined by core cancer team.
  Interventions: Other: questionnaire administration; Procedure: quality-of-life assessment
- DMP (experimental group): Patients undergo a systematic approach regarding specific domains related to their disease focusing on supportive care and symptom management determined by a multidisciplinary team of providers to help patients and caregivers manage.
  Interventions: Other: questionnaire administration; Procedure: quality-of-life assessment

INTERVENTIONS:
Other: questionnaire administration — Patients complete questionnaires.
Procedure: quality-of-life assessment — Patients undergo quality-of-life assessments.

SUMMARY:
RATIONALE: A disease management program may be more effective than standard therapy in improving quality of life and controlling symptoms in patients with cancer.

PURPOSE: This clinical trial is studying a disease management program to see how well it works compared with usual care in patients with stage III or stage IV lung cancer, stage III or stage IV pancreatic cancer, stage III or stage IV ovarian cancer, or stage III or stage IV colorectal cancer, and their caregivers.

DETAILED DESCRIPTION:
OBJECTIVES:

* To examine the effects of the expansion of the current disease-management program (DMP) in patients with stage III or IV lung pancreatic, ovarian, or colorectal cancer.
* To determine whether there is a difference in resource use (number of chemotherapy treatments in the last 30 days of life, number of emergency room visits, number of days of hospice and hospitalization) among patients who have participated in a DMP compared to those receiving usual care.
* To determine whether there is a difference in patient outcomes (health-related quality of life, spiritual well being, satisfaction with care) among patients who have participated in a DMP compared to those receiving usual care.
* To determine whether there is a difference in caregiver outcomes (mood state, satisfaction with care, satisfaction with end-of-life care, and burden of care giving) among caregivers of patients who have participated in a DMP compared to those receiving usual care.
* To determine whether differences in patient and caregiver outcomes remain after controlling for the influence of demographic, clinical, and organizational covariates.
* To determine the extent of differences in patient and caregiver outcomes achieved through improvements in collaboration and problem solving.

OUTLINE: Patients are stratified according to type of current supportive care (usual care vs comprehensive disease-management program [DMP]).

* Usual care (control group): Patients undergo usual care as determined by core cancer team.
* DMP (experimental group): Patients undergo a systematic approach regarding specific domains related to their disease, focusing on supportive care and symptom management determined by a multidisciplinary team of providers to help patients and caregivers manage.

Patients and caregivers are interviewed at baseline, 3, 9, and 15 months. Patients who transfer to hospice/palliative care treatment complete an additional questionnaire at the time of transfer and 3 weeks after transfer. If a patient death occurs during study, the caregiver is interviewed at 2 months after death.

Patient resource-use data is collected via billing data from hospital or clinic charts at the end of the patient's participation in the study and via monthly hospital and clinical chart review. Hospital visits, chemotherapy use, and hospice days are also measured as patient resource use.

Healthcare team members are interviewed weekly to measure contact time with patients. Team members receive team problem solving and team collaboration tools every 4 months for up to 37 months. Key members (nurse manager and physician clinical director) are also interviewed every 4 months.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically confirmed diagnosis of 1 of the following:

  * Lung cancer
  * Pancreatic cancer
  * Ovarian cancer
  * Colorectal cancer
* Stage III or IV disease
* Receiving care at the Ireland Cancer Center

PATIENT CHARACTERISTICS:

* ECOG performance status 0-3
* Life expectancy ≥ 3 months
* No cognitive impairment
* May not transfer care out of geographic area
* Must have caregiver available to participate

PRIOR CONCURRENT THERAPY:

* Not specified

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: primary care clinic
Sampling Method: Probability Sample
Enrollment: 605 (Actual)
Dates: Start 2007-08; Primary Completion 2011-12 (Actual); Study Completion 2011-12 (Actual)

PRIMARY OUTCOMES:
Patient resource use | at the end of the patient's participation in the study and via monthly hospital and clinical chart review.
Symptoms | Patients and caregivers are interviewed at baseline, 3, 9, and 15 months
Quality of life | Patients and caregivers are interviewed at baseline, 3, 9, and 15 months
Proportion of patients meeting expectations regarding care and treatment | Patients and caregivers are interviewed at baseline, 3, 9, and 15 months
Patient spiritual well-being | Patients and caregivers are interviewed at baseline, 3, 9, and 15 months
Caregiver mood state | Patients and caregivers are interviewed at baseline, 3, 9, and 15 months
Caregiver burden | Patients and caregivers are interviewed at baseline, 3, 9, and 15 months
Proportion of caregivers meeting expectations regarding care and treatment | Patients and caregivers are interviewed at baseline, 3, 9, and 15 months
Caregiver's satisfaction with end-of-life care | caregiver is interviewed at 2 months after death.

CONTACTS AND LOCATIONS:
Overall Officials: Barbara Daly, PhD, RN, Principal Investigator — Case Medical Center, University Hospitals Seidman Cancer Center, Case Comprehensive Cancer Center
Locations (1):
- Case Medical Center, University Hospitals Seidman Cancer Center, Case Comprehensive Cancer Center, Cleveland, Ohio, United States

REFERENCES:
- [Derived] Daly BJ, Douglas SL, Gunzler D, Lipson AR. Clinical trial of a supportive care team for patients with advanced cancer. J Pain Symptom Manage. 2013 Dec;46(6):775-84. doi: 10.1016/j.jpainsymman.2012.12.008. Epub 2013 Mar 22. PMID 23523362